CLINICAL TRIAL: NCT02908607
Title: Thermal Imaging for Cervical Cancer Screening and Early Detection
Brief Title: Thermal Imaging for Evaluation of the Cervix
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Yfat kadan, Dr., Meir Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0104-16-MMC
Record Dates: First submitted 2016-09-18; First posted 2016-09-21 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Cervical Neoplasia

ARMS (1):
- experimental (Experimental): 3 groups of patients will be participated: women with cancer, women with premalignant lesions and women with a normal cervix. All patients will undergo the same examination
  Interventions: Device: Thermal imaging

INTERVENTIONS:
Device: Thermal imaging — Examination of the cervix by thermal imaging camera

SUMMARY:
When screening results for cervical premalignant lesions are positive, colposcopy is recommended. This is highly sensitive screening method. However, specificity of the test is of low.

Thus, a technology that improves the accuracy of the colposcopic exam is needed.

This is a feasibility study with the goal of examining the performance of a thermal imaging camera in the detection of cervical malignant and premalignant lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18
* Women with premalignant cervical lesions who are candidates for conization (group A)
* Women with a normal cervix who are candidates for hysterectomy (group B)
* Women with newly diagnosed cervical cancer

Exclusion Criteria:

* For group A and B - women that had conization in the past

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-11; Primary Completion 2019-03 (Estimated)

PRIMARY OUTCOMES:
The rate of identification of premalignant and malignant lesions of the cervix by thermal imaging | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Meir medical center, Kfar Saba, Israel